CLINICAL TRIAL: NCT02990806
Title: A Randomized, Double-Blind, Multicenter, 3 Stage, Efficacy and Safety Study of NI-071 and US-Licensed Remicade® (Infliximab) for the Treatment of Patients With Rheumatoid Arthritis
Brief Title: A Phase 3 Study of NI-071 in Participants With Rheumatoid Arthritis (RADIANCE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nichi-Iko Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NI071F2
Record Dates: First submitted 2016-11-21; First posted 2016-12-13 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stages 1, 2 and 3: NI-071 Group (Experimental): Participants received intravenous (IV) infusion of NI-071 at a dose of 3 milligrams/kilograms (mg/kg) at Weeks 0, 2, 6, 14 during stage 1 and at Weeks 22, 30, 38, 46, and 54 during stage 2. Participants were followed up to Week 62 (Stage 3).
  Interventions: Drug: NI-071
- Stage 1: Remicade-US Group (Experimental): Participants received IV infusion of Remicade-US (infliximab) at a dose of 3 mg/kg at Weeks 0, 2, 6, 14 during stage 1.
  Interventions: Drug: Remicade
- Stage 2 and Stage 3: Remicade US to Remicade-US Group (Experimental): Participants who received Remicade US during stage 1; were re-randomized during stage 2 to continue Remicade-US dose 3 mg/kg from Week 22 through Week 54 with every 8 weeks dosing intervals. Participants were followed up to Week 62 (Stage 3).
  Interventions: Drug: Remicade
- Stage 2 and Stage 3: Remicade US to Switch Group (Experimental): Participants who received Remicade US during stage 1; were re-randomized during stage 2 and received IV infusion of NI-071 at Week 22 followed by Remicade-US at Week 30, followed by NI-071 at Weeks 38, 46, and 54. Participants were followed up to week 62 (Stage 3).
  Interventions: Drug: NI-071; Drug: Remicade

INTERVENTIONS:
Drug: NI-071 — IV infusion.
  Arms: Stage 2 and Stage 3: Remicade US to Switch Group; Stages 1, 2 and 3: NI-071 Group
Drug: Remicade — IV infusion.
  Arms: Stage 1: Remicade-US Group; Stage 2 and Stage 3: Remicade US to Remicade-US Group; Stage 2 and Stage 3: Remicade US to Switch Group

SUMMARY:
The purpose of this study was to demonstrate similarity of NI-071 (proposed biosimilar to infliximab) to US REMICADE® (reference product) in terms of safety and efficacy in participants with rheumatoid arthritis (RA) not adequately responding to methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of rheumatoid arthritis (RA) as defined by the 2010 American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) classification criteria.
* Patients have active RA, as confirmed by the following criteria:

  * ≥6 swollen joints and ≥6 tender joints at screening and baseline (28-joint count).
  * Either C-reactive protein (CRP) ≥0.7 mg/dL (≥7.0 mg/L) or erythrocyte sedimentation rate (ESR) ≥28 mm/h at screening.
* Patients taking methotrexate (MTX) (oral or parenteral) for at least 3 months prior to screening and at a stable dose of between 10 and 25 mg/week for at least 8 weeks. Concomitant folic/folinic acid at a dose of at least 5 mg/week is to be taken during the study; patients can start treatment with folic/folinic acid at screening if not already receiving it.
* If the patient is currently taking non-steroidal anti-inflammatory drugs (NSAIDs), the patient must be on a stable dose for at least 4 weeks prior to screening and during the study.
* Patients who are ≥18 and ≤75 years of age at screening.

Exclusion Criteria:

* Patients who are rated as Class IV according to the 1991 ACR revised criteria for classification of global functional status for RA.
* Patients who have received disease-modifying anti rheumatic drugs (DMARDs), other than MTX, within a period prior to screening shorter than the washout period appropriate to the pharmacodynamic profile of the specific drug.
* Patients who have received immunosuppressive drugs within 4 weeks prior to screening. Patients on a stable dose of oral corticosteroids (≤10 mg/day prednisone or equivalent) for ≥4 weeks prior to screening are permitted.
* Patients who have received intra-articular, intramuscular, intravenous, or epidural injection of corticosteroids within 4 weeks prior to screening.
* Patients who have received intra-articular sodium hyaluronate injections within 4 weeks prior to screening.
* Patients who have received surgical therapy for RA such as synovectomy or arthroplasty within 6 months prior to screening.
* Patients who have received arthrocentesis within 4 weeks prior to screening.
* Patients who have had prior treatment with infliximab.
* Patients who have had prior treatment with >1 biological drug or >1 protein kinase inhibitor for RA either as part of clinical management or during a clinical study.
* Patients who have had prior treatment with tumor necrosis factor alpha (TNF-α) inhibitors for RA who had lack of efficacy as per clinical judgment (primary failure). Patients who have discontinued TNF-α inhibitors for RA (other than infliximab) for any reason other than lack of efficacy are allowed.
* Presence of chronic or acute infection at screening, including positive result for active tuberculosis (TB).
* Patients with an acute infection requiring parenteral antibiotics within 4 weeks of study dosing or requiring oral/topical antibiotics within 2 weeks of study dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (98):
- United States (58):
  - Nichi-Iko Investigational Site, Little Rock, Arkansas
  - Nichi-Iko Investigational Site, Los Angeles, California
  - Nichi-Iko Investigational Site, Ventura, California
  - Nichi-Iko Investigational Site, Whittier, California
  - Nichi-Iko Investigational Site, Hamden, Connecticut
  - Nichi-Iko Investigational Site, Boca Raton, Florida
  - Nichi-Iko Investigational Site, Boynton Beach, Florida
  - Nichi-Iko Investigational Site, Brandon, Florida
  - Nichi-Iko Investigational Site, Doral, Florida
  - Nichi-Iko Investigational Site, Hialeah, Florida
  - Nichi-Iko Investigational Site, Jacksonville, Florida
  - Nichi-Iko Investigational Site, Miami, Florida
  - Nichi-Iko Investigational Site, Miami Lakes, Florida
  - Nichi-Iko Investigational Site, Pembroke Pines, Florida
  - Nichi-Iko Investigational Site, Pinellas Park, Florida
  - Nichi-Iko Investigational Site, Sarasota, Florida
  - Nichi-Iko Investigational Site, West Palm Beach, Florida
  - Nichi-Iko Investigational Site, Decatur, Georgia
  - Nichi-Iko Investigational Site, Meridian, Idaho
  - Nichi-Iko Investigational Site, Lexington, Kentucky
  - Nichi-Iko Investigational Site, Louisville, Kentucky
  - Nichi-Iko Investigational Site, Worcester, Massachusetts
  - Nichi-Iko Investigational Site, Ann Arbor, Michigan
  - Nichi-Iko Investigational Site, Grand Rapids, Michigan
  - Nichi-Iko Investigational Site, Lansing, Michigan
  - Nichi-Iko Investigational Site, Tupelo, Mississippi
  - Nichi-Iko Investigational Site, Las Vegas, Nevada
  - Nichi-Iko Investigational Site, Freehold, New Jersey
  - Nichi-Iko Investigational Site, Durham, North Carolina
  - Nichi-Iko Investigational Site, Greenville, North Carolina
  - Nichi-Iko Investigational Site, Salisbury, North Carolina
  - Nichi-Iko Investigational Site, Wilmington, North Carolina
  - Nichi-Iko Investigational Site, Cincinnati, Ohio
  - Nichi-Iko Investigational Site, Columbus, Ohio
  - Nichi-Iko Investigational Site, Middleburg Heights, Ohio
  - Nichi-Iko Investigational Site, Oklahoma City, Oklahoma
  - Nichi-Iko Investigational Site, Duncansville, Pennsylvania
  - Nichi-Iko Investigational Site, Media, Pennsylvania
  - Nichi-Iko Investigational Site, Wyomissing, Pennsylvania
  - Nichi-Iko Investigational Site, Charleston, South Carolina
  - Nichi-Iko Investigational Site, Fort Mill, South Carolina
  - Nichi-Iko Investigational Site, Jackson, Tennessee
  - Nichi-Iko Investigational Site, Memphis, Tennessee
  - Nichi-Iko Investigational Site, Amarillo, Texas
  - Nichi-Iko Investigational Site, Baytown, Texas
  - Nichi-Iko Investigational Site, Beaumont, Texas
  - Nichi-Iko Investigational Site, Corpus Christi, Texas
  - Nichi-Iko Investigational Site, Cypress, Texas
  - Nichi-Iko Investigational Site, El Paso, Texas
  - Nichi-Iko Investigational Site, Galveston, Texas
  - Nichi-Iko Investigational Site, Houston, Texas
  - Nichi-Iko Investigational Site, Mesquite, Texas
  - Nichi-Iko Investigational Site, Nassau Bay, Texas
  - Nichi-Iko Investigational Site, San Antonio, Texas
  - Nichi-Iko Investigational Site, Sugar Land, Texas
  - Nichi-Iko Investigational Site, Tomball, Texas
  - Nichi-Iko Investigational Site, Webster, Texas
  - Nichi-Iko Investigational Site, Chesapeake, Virginia
- Czechia (4):
  - Nichi-Iko Investigational Site, Ostrava
  - Nichi-Iko Investigational Site, Prague
  - Nichi-Iko Investigational Site, Uherské Hradišté
  - Nichi-Iko Investigational Site, Zlín
- Poland (8):
  - Nichi-Iko Investigational Site, Bialystok
  - Nichi-Iko Investigational Site, Katowice
  - Nichi-Iko Investigational Site, Lodz
  - Nichi-Iko Investigational Site, Lublin
  - Nichi-Iko Investigational Site, Olsztyn
  - Nichi-Iko Investigational Site, Poznan
  - Nichi-Iko Investigational Site, Torun
  - Nichi-Iko Investigational Site, Warsaw
- Puerto Rico (2):
  - Nichi-Iko Investigational Site, Caguas
  - Nichi-Iko Investigational Site, San Juan
- Russia (10):
  - Nichi-Iko Investigational Site, Kemerovo
  - Nichi-Iko Investigational Site, Moscow
  - Nichi-Iko Investigational Site, Novosibirsk
  - Nichi-Iko Investigational Site, Penza
  - Nichi-Iko Investigational Site, Petrozavodsk
  - Nichi-Iko Investigational Site, Ryazan
  - Nichi-Iko Investigational Site, Saint Petersburg
  - Nichi-Iko Investigational Site, Tomsk
  - Nichi-Iko Investigational Site, Vladimir
  - Nichi-Iko Investigational Site, Yaroslavl
- Spain (4):
  - Nichi-Iko Investigational Site, A Coruña
  - Nichi-Iko Investigational Site, Barcelona
  - Nichi-Iko Investigational Site, Santiago de Compostela
  - Nichi-Iko Investigational Site, Seville
- Ukraine (8):
  - Nichi-Iko Investigational Site, Kharkiv
  - Nichi-Iko Investigational Site, Kyiv
  - Nichi-Iko Investigational Site, Lviv
  - Nichi-Iko Investigational Site, Odesa
  - Nichi-Iko Investigational Site, Ternopil
  - Nichi-Iko Investigational Site, Vinnytsia
  - Nichi-Iko Investigational Site, Zaporizhzhya
  - Nichi-Iko Investigational Site, Zhytomyr
- United Kingdom (4):
  - Nichi-Iko Investigational Site, Bury St Edmunds
  - Nichi-Iko Investigational Site, Gillingham
  - Nichi-Iko Investigational Site, Leicester
  - Nichi-Iko Investigational Site, Truro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 97 investigative site in Czech Republic, Poland, Russia, Spain, Ukraine, and the United States in the study from 19 January 2017 to 20 May 2019.
Pre-assignment Details: The study consisted of 3 stages: the biosimilarity stage (Stage 1), the interchangeability stage (Stage 2), and the safety follow-up stage (Stage 3). A total of 683 participants were randomized in a 2:1 ratio to the Remicade-US and NI-071 groups during Stage 1. In Stage 2 participants in the original Remicade-US group were re-randomized (1:1) to a Remicade-US group and a Switch group (to assess the effects of switching between Remicade-US and NI-071).
Groups:
- Stage 1 and 2: NI-071 Group: Participants received intravenous (IV) infusion of NI-071 at a dose of 3 milligrams/kilograms (mg/kg) at Weeks 0, 2, 6, 14 during stage 1 and at Weeks 22, 30, 38, 46, and 54 during stage 2. Participants were followed up to Week 62 during safety follow-up.
Period: Stage 1 (22 Weeks)
Arm/Group | Stage 1 and 2: NI-071 Group | Stage 1: Remicade-US Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Started | 228 | 455 (Participants randomized to receive Remicade-US during stage 1.) | 0 | 0
Safety Population | 227 | 451 | 0 | 0
Completed | 214 | 399 | 0 | 0
Not Completed | 14 | 56 | 0 | 0
Not completed — Adverse Event | 1 | 15 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Initiated protocol-prohibited medication | 2 | 2 | 0 | 0
Not completed — Noncompliant with visit schedule and/or protocol | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 26 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Required antibiotics resulting in drug interruption >2 weeks | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0
Not completed — Other | 1 | 3 | 0 | 0
Period: Stage 2 (32 Weeks)
Arm/Group | Stage 1 and 2: NI-071 Group | Stage 1: Remicade-US Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Started | 214 | 0 | 201 (399 participants completed stage 1 of Remicade US group, of which 201 participants were randomized to this arm.) | 196 (399 participants completed stage 1 of Remicade US group, of which 196 participants were randomized to this arm.)
Completed | 172 | 0 | 173 | 162
Not Completed | 42 | 0 | 28 | 34
Not completed — Adverse Event | 9 | 0 | 7 | 7
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 1 | 0
Not completed — Diagnosed with malignancy | 1 | 0 | 0 | 1
Not completed — Required antibiotics resulting in drug interruption | 1 | 0 | 1 | 1
Not completed — Initiated protocol-prohibited medication | 1 | 0 | 0 | 2
Not completed — Noncompliant with visit schedule and/or protocol | 2 | 0 | 6 | 5
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2
Not completed — Protocol deviation | 2 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 14 | 0 | 4 | 8
Not completed — Lack of Efficacy | 4 | 0 | 2 | 3
Not completed — Other | 3 | 0 | 4 | 1
Not completed — Ineligible according to Tuberculosis (TB) criteria | 0 | 0 | 0 | 1
Period: Stage 3 (Safety Follow-up) (8 Weeks)
Arm/Group | Stage 1 and 2: NI-071 Group | Stage 1: Remicade-US Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Started | 172 | 0 | 173 | 162
Completed | 163 | 0 | 162 | 152
Not Completed | 9 | 0 | 11 | 10
Not completed — Adverse Event | 5 | 0 | 4 | 3
Not completed — Physician Decision | 1 | 0 | 1 | 1
Not completed — Noncompliant with visit schedule and/or protocol | 2 | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 2
Not completed — Initiated protocol-prohibited medication | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were randomized, irrespective of any deviation from the protocol or premature discontinuation.
Groups:
- Stage 1: NI-071 Group: Participants received intravenous (IV) infusion of NI-071 at a dose of 3 milligrams/kilograms (mg/kg) at Weeks 0, 2, 6, 14 during stage 1.
- Total: Total of all reporting groups
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group | Total
Number analyzed (Participants) | 228 | 455 | 683
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.0) | 53.7 (11.9) | 53.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 372 | 545
  Male | 55 | 83 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 103 | 153
  Not Hispanic or Latino | 174 | 350 | 524
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 25 | 42
  White | 211 | 424 | 635
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants Who Achieved 20 Percent (%) American College of Rheumatology C-reactive Protein (ACR20-CRP) Response Rate at Week 22
Description: ACR20 was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 20% improvement from baseline in the tender/painful joint count. ii) A 20% improvement from baseline in the swollen joint count. iii) A 20% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity visual analog scale (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS) (0= no symptoms;100=severe symptoms), c) Participant pain assessment (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), d) Health Assessment Questionnaire-Disability Index (HAQ-DI), total score ranging from 0-3 with lower scores meaning less disability, e) CRP.
Time Frame: At Week 22
Population: The Intent to Treat (ITT) included all participants who were randomized, irrespective of any deviation from the protocol or premature discontinuation. Data for this outcome measure was planned to be collected and analyzed for Stage 1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Stage 1: NI-071 Group: Participants received IV infusion of NI-071 at a dose of 3 mg/kg at Weeks 0, 2, 6, 14 during stage 1.
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 228 | 455
percentage of participants | 56.6 [50.1 to 63.0] | 53.0 [48.4 to 57.6]
Statistical Analysis 1: Comparison: Stage 1: NI-071 Group vs Stage 1: Remicade-US Group; Test type: Equivalence — A test for equivalence was carried out using an asymmetric margin (-12%, 15%) pre-specified in protocol and a two 1-sided test (TOST) analysis with α=0.05 for each 1-sided statistical test; Percentage difference = 3.6, 95% CI 2-sided [-4.3 to 11.5], Standard Error of Mean 0.04

2. Primary Outcome: Stage 2 and 3: Area Under the Serum Concentration-time Curve Interval (AUCtau) of NI-071 and Remicade US
Description: AUCtau of NI-071 and Remicade US in stage 2 and 3 was reported. As this was an interchangeability study, the NI-071 and Remicade only were the comparators and then switch study showed same measurement in relationship to the non-switched participants. Hence, combined data was assessed and collected in participants from Remicade US to Switch Group.
Time Frame: Week 46: Pre-dose, 1 hour after infusion, at end of infusion, at 4 hours and 24 hours after infusion and at Week 47, Week 48, Week 50, Week 52, and Week 54 post-dose
Population: Pharmacokinetic (PK) population included all participants in the full analysis set (FAS) in Stage 1 who have valid PK assessments through Stage 2. The FAS included all participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR20 efficacy assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Stage 1.
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (h*ng/mL)
Groups:
- Stage 2 and Stage 3: NI-071 Group: Participants received IV infusion of NI-071 at a dose of 3 mg/kg at Weeks 22, 30, 38, 46, and 54 during stage 2. Participants were followed up to Week 62 (Stage 3).
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 149 | 146 | 135
hour*nanograms per milliliter (h*ng/mL) | 12949622.78 (6999387.76) | 12859923.90 (8228379.79) | 12040415.23 (6624933.11)

3. Primary Outcome: Stage 2 and 3: Maximum Observed Serum Concentration (Cmax) of NI-071 and Remicade US
Description: Cmax of NI-071 and Remicade US was reported. As this was an interchangeability study, the NI-071 and Remicade only were the comparators and then switch study showed same measurement in relationship to the non-switched participants. Hence, combined data was assessed and collected in participants from Remicade US to Switch Group.
Time Frame: as for outcome 2
Population: PK population included all participants in the FAS in Stage 1 who have valid PK assessments through Stage 2. The FAS included all participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR20 efficacy assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for Stage 1.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 159 | 155 | 146
nanograms per milliliter (ng/mL) | 66298.1 (21756.8) | 63649.0 (16566.2) | 61660.8 (18696.5)

4. Secondary Outcome: Stage 1: Change From Baseline in the Disease Activity Score Based on 28 Joints (DAS28) C-reactive Protein (CRP) at Weeks 2, 6, 14, 18, and 22
Description: The DAS28-CRP was a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints [assessed on 2-point scale (0=absent; 1=present]), swollen joint count (out of 28 evaluated joints[assessed on 2-point scale (0=absent; 1=present)]), Participant's global assessment of disease activity (assessed on 0-100 mm VAS; where higher scores denotes severe symptoms), and high-sensitivity C-reactive protein (hsCRP; in mg/L). Total Scores on the DAS28-CRP range from 0 to approximately 10 (0=very good, no symptoms; 10=very poor, severe symptoms), where higher scores indicate more disease activity. A negative change from baseline indicates improvement in disease activity.
Time Frame: Baseline, Weeks 2, 6, 14, 18, and 22
Population: The FAS population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR20 efficacy assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
score on a scale
  Baseline | 5.816 (0.822) | 5.898 (0.787)
  Change at Week 2: number analyzed (Participants) | 226 | 443
  Change at Week 2 | -1.094 (0.881) | -1.169 (0.931)
  Change at Week 6: number analyzed (Participants) | 224 | 441
  Change at Week 6 | -1.542 (1.041) | -1.650 (1.114)
  Change at Week 14: number analyzed (Participants) | 218 | 423
  Change at Week 14 | -1.828 (1.137) | -1.812 (1.221)
  Change at Week 18: number analyzed (Participants) | 215 | 407
  Change at Week 18 | -2.070 (1.159) | -2.156 (1.193)
  Change at Week 22: number analyzed (Participants) | 217 | 404
  Change at Week 22 | -1.835 (1.247) | -1.978 (1.209)

5. Secondary Outcome: Stage 2 and 3: Change From Baseline in the Disease Activity Score Based on 28 Joints (DAS28) C-reactive Protein (CRP) at Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Description: as for outcome 4
Time Frame: Baseline, Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stage 2 and Stage 3: NI-071 Group: Participants from Stage 1 continued to receive IV infusion of NI-071 at a dose of 3 mg/kg at Weeks 22, 30, 38, 46, and 54 during Stage 2. Participants were followed up to Week 62 (Stage 3).
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 212 | 198 | 194
score on a scale
  Change at Week 26 | -2.199 (1.238) | -2.317 (1.227) | -2.192 (1.180)
  Change at Week 30: number analyzed (Participants) | 203 | 189 | 188
  Change at Week 30 | -2.106 (1.269) | -2.298 (1.251) | -2.092 (1.230)
  Change at Week 34: number analyzed (Participants) | 199 | 182 | 184
  Change at Week 34 | -2.379 (1.251) | -2.586 (1.187) | -2.446 (1.266)
  Change at Week 38: number analyzed (Participants) | 190 | 183 | 173
  Change at Week 38 | -2.281 (1.234) | -2.331 (1.258) | -2.321 (1.376)
  Change at Week 42: number analyzed (Participants) | 182 | 181 | 171
  Change at Week 42 | -2.415 (1.228) | -2.630 (1.226) | -2.519 (1.236)
  Change at Week 46: number analyzed (Participants) | 173 | 176 | 164
  Change at Week 46 | -2.242 (1.203) | -2.387 (1.270) | -2.207 (1.217)
  Change at Week 50: number analyzed (Participants) | 174 | 171 | 162
  Change at Week 50 | -2.444 (1.156) | -2.679 (1.245) | -2.551 (1.172)
  Change at Week 54: number analyzed (Participants) | 167 | 165 | 162
  Change at Week 54 | -2.443 (1.212) | -2.462 (1.189) | -2.247 (1.298)
  Change at Week 58: number analyzed (Participants) | 165 | 162 | 155
  Change at Week 58 | -2.568 (1.211) | -2.739 (1.236) | -2.450 (1.227)
  Change at Week 62: number analyzed (Participants) | 162 | 161 | 154
  Change at Week 62 | -2.466 (1.238) | -2.605 (1.276) | -2.404 (1.327)

6. Secondary Outcome: Stage 1: Change From Baseline in the Disease Activity Score Based on 28 Joints (DAS28)-Erythrocyte Sedimentation Rate (ESR) at Weeks 2, 6, 14, 18, and 22
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. The components of the DAS28 (ESR) assessment included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (millimeters per hour) and GH recorded on 100mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). DAS28 (ESR) was calculated as 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*ln(ESR [mm/hour] + 0.014*GH [mm]; where, TJC28 = number of painful joints out of 28 joints, SJC28 = number of swollen joints out of 28 joints, GH = score of the participant global assessment of disease activity, ln = natural logarithm, sqrt = square root of. Total score range: 0 to 9.4, higher score indicated more disease activity. A negative change from baseline indicates improvement in disease activity.
Time Frame: Baseline, Weeks 2, 6, 14, 18, and 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 445
score on a scale
  Baseline | 6.552 (0.861) | 6.655 (0.755)
  Change at Week 2: number analyzed (Participants) | 225 | 442
  Change at Week 2 | -1.060 (0.915) | -1.161 (0.893)
  Change at Week 6: number analyzed (Participants) | 224 | 437
  Change at Week 6 | -1.588 (1.112) | -1.778 (1.174)
  Change at Week 14: number analyzed (Participants) | 216 | 420
  Change at Week 14 | -2.002 (1.254) | -1.951 (1.266)
  Change at Week 18: number analyzed (Participants) | 215 | 406
  Change at Week 18 | -2.291 (1.300) | -2.345 (1.278)
  Change at Week 22: number analyzed (Participants) | 217 | 402
  Change at Week 22 | -2.060 (1.386) | -2.195 (1.326)

7. Secondary Outcome: Stage 2 and 3: Change From Baseline in the Disease Activity Score Based on 28 Joints (DAS28)-Erythrocyte Sedimentation Rate (ESR) at Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Description: DAS28 is a measure of disease activity in participants with rheumatoid arthritis, derived using differential weighting given to each of the four components. The components of the DAS28 (ESR) assessment included: TJC with 28 joints assessed, SJC with 28 joints assessed, ESR (millimeters per hour) and Patient Global Assessment (PtGA) recorded on 100mm VAS (0=very good, no symptoms;100=very poor, severe symptoms). DAS28 (ESR) was calculated as 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.70*ln(ESR [mm/hour] + 0.014*GH [mm]; where, TJC28 = number of painful joints out of 28 joints, SJC28 = number of swollen joints out of 28 joints, GH = score of the participant global assessment of disease activity, ln = natural logarithm, sqrt = square root of. Total score range: 0 to 9.4, higher score indicated more disease activity. A negative change from baseline indicates improvement in disease activity.
Time Frame: Baseline, Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Stage 2 and Stage 3: Remicade US to Switch Group: Participants who received Remicade US during stage 1; were re-randomized during stage 2 received IV infusion of NI-071 at Week 22 followed by Remicade-US at Week 30, followed by NI-071 at Weeks 38, 46, and 54. Participants were followed up to week 62 (Stage 3).
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 212 | 198 | 193
score on a scale
  Change at Week 26 | -2.387 (1.393) | -2.533 (1.395) | -2.375 (1.304)
  Change at Week 30: number analyzed (Participants) | 201 | 189 | 187
  Change at Week 30 | -2.346 (1.457) | -2.533 (1.349) | -2.261 (1.374)
  Change at Week 34: number analyzed (Participants) | 199 | 182 | 183
  Change at Week 34 | -2.602 (1.416) | -2.864 (1.303) | -2.609 (1.376)
  Change at Week 38: number analyzed (Participants) | 190 | 183 | 172
  Change at Week 38 | -2.516 (1.478) | -2.535 (1.314) | -2.493 (1.518)
  Change at Week 42: number analyzed (Participants) | 182 | 181 | 170
  Change at Week 42 | -2.650 (1.372) | -2.847 (1.258) | -2.691 (1.433)
  Change at Week 46: number analyzed (Participants) | 173 | 175 | 163
  Change at Week 46 | -2.494 (1.352) | -2.625 (1.322) | -2.406 (1.364)
  Change at Week 50: number analyzed (Participants) | 174 | 171 | 161
  Change at Week 50 | -2.649 (1.291) | -2.964 (1.302) | -2.708 (1.303)
  Change at Week 54: number analyzed (Participants) | 167 | 165 | 161
  Change at Week 54 | -2.619 (1.385) | -2.662 (1.221) | -2.403 (1.410)
  Change at Week 58: number analyzed (Participants) | 165 | 162 | 154
  Change at Week 58 | -2.764 (1.385) | -2.985 (1.337) | -2.617 (1.376)
  Change at Week 62: number analyzed (Participants) | 162 | 161 | 153
  Change at Week 62 | -2.663 (1.439) | -2.864 (1.371) | -2.574 (1.470)

8. Secondary Outcome: Stage 1: Percentage of Participants Who Achieved 20 Percent (%) American College of Rheumatology C-reactive Protein (ACR-CRP) Response Rate
Description: ACR20 was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 20% improvement from baseline in the tender/painful joint count. ii) A 20% improvement from baseline in the swollen joint count. iii) A 20% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3 with lower scores meaning less disability, e) CRP.
Time Frame: At Weeks 2, 6, 14, 18, and 22
Population: The FAS population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR20 efficacy assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure. Last observation carried forward (LOCF) method was used to carry forward any of the individually missing component values, and from that mix of actual and carried-forward values, the ACR responder status was determined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
percentage of participants
  At Week 2 | 31.3 [25.2 to 37.3] | 32.5 [28.2 to 36.9]
  At Week 6 | 47.1 [40.6 to 53.6] | 54.3 [49.6 to 58.9]
  At Week 14 | 56.4 [49.9 to 62.8] | 51.1 [46.5 to 55.8]
  At Week 18 | 62.6 [56.3 to 68.9] | 61.7 [57.1 to 66.2]
  At Week 22 | 56.8 [50.4 to 63.3] | 54.5 [49.9 to 59.1]

9. Secondary Outcome: Stage 2 and 3: Percentage of Participants Who Achieved 20 Percent (%) American College of Rheumatology C-reactive Protein (ACR-CRP) Response Rate
Description: ACR20 was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 20% improvement from baseline in the tender/painful joint count. ii) A 20% improvement from baseline in the swollen joint count. iii) A 20% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3 with lower scores meaning less disability, e) CRP.
Time Frame: At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: Full Analysis Set population included participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR20 efficacy assessment. Overall Number of Participants indicates the number of patients with FAS. The patient number of FAS is the number of patients evaluated at baseline, which is different from number of patients who started Stage 2 or 3. ACR 20 (CRP) response rate/visit was calculated based on the number of patients achieving ACR20 criteria divided by FAS number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 248 | 197
percentage of participants
  At Week 26 | 62.6 [56.3 to 68.9] | 56.5 [50.3 to 62.6] | 61.9 [55.1 to 68.7]
  At Week 30 | 55.5 [49.0 to 62.0] | 48.8 [42.6 to 55.0] | 57.9 [51.0 to 64.8]
  At Week 34 | 61.7 [55.3 to 68.0] | 55.6 [49.5 to 61.8] | 61.4 [54.6 to 68.2]
  At Week 38 | 52.0 [45.5 to 58.5] | 47.6 [41.4 to 53.8] | 57.9 [51.0 to 64.8]
  At Week 42 | 54.6 [48.1 to 61.1] | 53.6 [47.4 to 59.8] | 59.4 [52.5 to 66.2]
  At Week 46 | 51.1 [44.6 to 57.6] | 48.0 [41.8 to 54.2] | 51.3 [44.3 to 58.2]
  At Week 50 | 54.2 [47.7 to 60.7] | 50.0 [43.8 to 56.2] | 59.9 [53.1 to 66.7]
  At Week 54 | 52.4 [45.9 to 58.9] | 47.2 [41.0 to 53.4] | 49.2 [42.3 to 56.2]
  At Week 58 | 52.4 [45.9 to 58.9] | 46.4 [40.2 to 52.6] | 56.9 [49.9 to 63.8]
  At Week 62 | 52.0 [45.5 to 58.5] | 46.4 [40.2 to 52.6] | 55.3 [48.4 to 62.3]

10. Secondary Outcome: Stage 1: Percentage of Participants Who Achieved Greater Than or Equal to (>=) 20% American College of Rheumatology (ACR20) Response Using Erythrocyte Sedimentation Rate (ESR)
Description: ACR20-ESR was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 20% improvement from baseline in the tender/painful joint count. ii) A 20% improvement from baseline in the swollen joint count. iii) A 20% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3 with lower scores meaning less disability, e) erythrocyte sedimentation rate (ESR).
Time Frame: At Weeks 2, 6, 14, 18, and 22
Population: The FAS population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR20 efficacy assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure. LOCF method was used to carry forward any of the individually missing component values, and from that mix of actual and carried-forward values, the ACR responder status was determined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
percentage of participants
  At Week 2 | 29.1 [23.2 to 35.0] | 31.8 [27.5 to 36.2]
  At Week 6 | 46.7 [40.2 to 53.2] | 54.3 [49.6 to 58.9]
  At Week 14 | 56.8 [50.4 to 63.3] | 52.2 [47.6 to 56.9]
  At Week 18 | 62.6 [56.3 to 68.9] | 62.3 [57.8 to 66.8]
  At Week 22 | 55.9 [49.5 to 62.4] | 56.3 [51.7 to 60.9]

11. Secondary Outcome: Stage 2 and 3: Percentage of Participants Who Achieved Greater Than or Equal to (>=) 20% American College of Rheumatology (ACR20) Response Using Erythrocyte Sedimentation Rate (ESR)
Description: ACR20-ESR was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 20% improvement from baseline in the tender/painful joint count. ii) A 20% improvement from baseline in the swollen joint count. iii) A 20% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3 with lower scores meaning less disability, e) (ESR.
Time Frame: At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 248 | 197
percentage of participants
  At Week 26 | 60.8 [54.4 to 67.1] | 55.6 [49.5 to 61.8] | 62.4 [55.7 to 69.2]
  At Week 30 | 58.1 [51.7 to 64.6] | 50.0 [43.8 to 56.2] | 57.4 [50.5 to 64.3]
  At Week 34 | 62.1 [55.8 to 68.4] | 56.9 [50.7 to 63.0] | 61.4 [54.6 to 68.2]
  At Week 38 | 56.4 [49.9 to 62.8] | 48.8 [42.6 to 55.0] | 59.4 [52.5 to 66.2]
  At Week 42 | 57.3 [50.8 to 63.7] | 54.4 [48.2 to 60.6] | 60.9 [54.1 to 67.7]
  At Week 46 | 53.7 [47.3 to 60.2] | 50.0 [43.8 to 56.2] | 54.3 [47.4 to 61.3]
  At Week 50 | 56.4 [49.9 to 62.8] | 50.8 [44.6 to 57.0] | 59.4 [52.5 to 66.2]
  At Week 54 | 54.6 [48.1 to 61.1] | 47.2 [41.0 to 53.4] | 50.8 [43.8 to 57.7]
  At Week 58 | 54.2 [47.7 to 60.7] | 48.8 [42.6 to 55.0] | 55.8 [48.9 to 62.8]
  At Week 62 | 52.4 [45.9 to 58.9] | 47.2 [41.0 to 53.4] | 54.3 [47.4 to 61.3]

12. Secondary Outcome: Stage 1: Percentage of Participants Who Achieved >=50% American College of Rheumatology C-reactive Protein (ACR50-CRP) Response Rate
Description: ACR50 was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 50% improvement from baseline in the tender/painful joint count. ii) A 50% improvement from baseline in the swollen joint count. iii) A 50% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3, with lower scores meaning less disability, e) CRP.
Time Frame: At Weeks 2, 6, 14, 18, and 22
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
percentage of participants
  At Week 2 | 8.4 [4.8 to 12.0] | 8.3 [5.7 to 10.9]
  At Week 6 | 16.3 [11.5 to 21.1] | 19.1 [15.4 to 22.7]
  At Week 14 | 24.7 [19.1 to 30.3] | 21.3 [17.5 to 25.1]
  At Week 18 | 32.2 [26.1 to 38.2] | 30.9 [26.7 to 35.2]
  At Week 22 | 27.8 [21.9 to 33.6] | 25.6 [21.5 to 29.6]

13. Secondary Outcome: Stage 2 and 3: Percentage of Participants Who Achieved >=50% American College of Rheumatology C-reactive Protein (ACR50-CRP) Response Rate
Description: as for outcome 12
Time Frame: At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: Full Analysis Set population included participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR50 efficacy assessment. Overall Number of Participants indicates the number of patients with FAS. The patient number of FAS is the number of patients evaluated at baseline, which is different from number of patients who started Stage 2 or 3. ACR 50 (CRP) response rate/visit was calculated based on the number of patients achieving ACR50 criteria divided by FAS number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 248 | 446
percentage of participants
  At Week 26 | 34.4 [28.2 to 40.5] | 32.3 [26.4 to 38.1] | 31.0 [24.5 to 37.4]
  At Week 30 | 30.0 [24.0 to 35.9] | 28.6 [23.0 to 34.3] | 29.4 [23.1 to 35.8]
  At Week 34 | 35.2 [29.0 to 41.5] | 34.3 [28.4 to 40.2] | 39.1 [32.3 to 45.9]
  At Week 38 | 31.3 [25.2 to 37.3] | 30.2 [24.5 to 36.0] | 34.0 [27.4 to 40.6]
  At Week 42 | 33.5 [27.3 to 39.6] | 36.7 [30.7 to 42.7] | 40.6 [33.8 to 47.5]
  At Week 46 | 30.8 [24.8 to 36.8] | 31.5 [25.7 to 37.2] | 30.5 [24.0 to 36.9]
  At Week 50 | 37.0 [30.7 to 43.3] | 34.7 [28.8 to 40.6] | 35.5 [28.8 to 42.2]
  At Week 54 | 36.6 [30.3 to 42.8] | 28.6 [23.0 to 34.3] | 32.5 [25.9 to 39.0]
  At Week 58 | 32.6 [26.5 to 38.7] | 32.7 [26.8 to 38.5] | 34.0 [27.4 to 40.6]
  At Week 62 | 30.8 [24.8 to 36.8] | 32.7 [26.8 to 38.5] | 28.4 [22.1 to 34.7]

14. Secondary Outcome: Stage 1: Percentage of Participants Who Achieved >=50% American College of Rheumatology (ACR50) Response Using ESR
Description: ACR50-ESR was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 50% improvement from baseline in the tender/painful joint count. ii) A 50% improvement from baseline in the swollen joint count. iii) A 50% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3, with lower scores meaning less disability, e) ESR.
Time Frame: At Weeks 2, 6, 14, 18, and 22
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
percentage of participants
  At Week 2 | 6.6 [3.4 to 9.8] | 6.7 [4.4 to 9.1]
  At Week 6 | 14.5 [10.0 to 19.1] | 17.9 [14.4 to 21.5]
  At Week 14 | 23.3 [17.8 to 28.9] | 21.7 [17.9 to 25.6]
  At Week 18 | 31.7 [25.7 to 37.8] | 29.6 [25.4 to 33.8]
  At Week 22 | 27.8 [21.9 to 33.6] | 26.7 [22.6 to 30.8]

15. Secondary Outcome: Stage 2 and Stage 3: Percentage of Participants Who Achieved >=50% American College of Rheumatology (ACR50) Response Using ESR
Description: as for outcome 14
Time Frame: At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 248 | 197
percentage of participants
  At Week 26 | 33.0 [26.9 to 39.2] | 31.9 [26.1 to 37.7] | 30.5 [24.0 to 36.9]
  At Week 30 | 29.1 [23.2 to 35.0] | 28.2 [22.6 to 33.8] | 28.4 [22.1 to 34.7]
  At Week 34 | 35.2 [29.0 to 41.5] | 34.7 [28.8 to 40.6] | 39.1 [32.3 to 45.9]
  At Week 38 | 32.2 [26.1 to 38.2] | 30.6 [24.9 to 36.4] | 32.5 [25.9 to 39.0]
  At Week 42 | 33.5 [27.3 to 39.6] | 36.7 [30.7 to 42.7] | 37.1 [30.3 to 43.8]
  At Week 46 | 29.5 [23.6 to 35.4] | 31.5 [25.7 to 37.2] | 29.4 [23.1 to 35.8]
  At Week 50 | 34.8 [28.6 to 41.0] | 34.3 [28.4 to 40.2] | 34.5 [27.9 to 41.2]
  At Week 54 | 36.1 [29.9 to 42.4] | 28.6 [23.0 to 34.3] | 29.4 [23.1 to 35.8]
  At Week 58 | 32.6 [26.5 to 38.7] | 32.3 [26.4 to 38.1] | 33.5 [26.9 to 40.1]
  At Week 62 | 29.1 [23.2 to 35.0] | 32.7 [26.8 to 38.5] | 27.9 [21.7 to 34.2]

16. Secondary Outcome: Stage 1: Percentage of Participants Who Achieved >=70% American College of Rheumatology C-reactive Protein (ACR70-CRP) Response Rate
Description: ACR70 was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 50% improvement from baseline in the tender/painful joint count. ii) A 70% improvement from baseline in the swollen joint count. iii) A 70% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3, with lower scores meaning less disability, e) CRP.
Time Frame: At Weeks 2, 6, 14, 18, and 22
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
percentage of participants
  At Week 2 | 0.9 [0.0 to 2.1] | 1.3 [0.3 to 2.4]
  At Week 6 | 6.6 [3.4 to 9.8] | 7.2 [4.8 to 9.6]
  At Week 14 | 11.0 [6.9 to 15.1] | 7.8 [5.4 to 10.3]
  At Week 18 | 15.0 [10.3 to 19.6] | 11.7 [8.7 to 14.6]
  At Week 22 | 10.6 [6.6 to 14.6] | 12.1 [9.1 to 15.1]

17. Secondary Outcome: Stage 2 and 3: Percentage of Participants Who Achieved >=70% American College of Rheumatology C-reactive Protein (ACR70-CRP) Response Rate
Description: ACR70 was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 50% improvement from baseline in the tender/painful joint count. ii) A 70% improvement from baseline in the swollen joint count. iii) A 70% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity VAS) (0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3, with lower scores meaning less disability, e) CRP.
Time Frame: At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: Full Analysis Set population included participants who received at least 1 dose of study drug and had at least 1 post-baseline ACR70 efficacy assessment. Overall Number of Participants indicates the number of patients with FAS. The patient number of FAS is the number of patients evaluated at baseline, which is different from number of patients who started Stage 2 or 3. ACR 70 (CRP) response rate/visit was calculated based on the number of patients achieving ACR70 criteria divided by FAS number.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 248 | 197
percentage of participants
  At Week 26 | 16.3 [11.5 to 21.1] | 14.5 [10.1 to 18.9] | 13.2 [8.5 to 17.9]
  At Week 30 | 16.3 [11.5 to 21.1] | 15.3 [10.8 to 19.8] | 13.2 [8.5 to 17.9]
  At Week 34 | 18.1 [13.1 to 23.1] | 18.1 [13.3 to 22.9] | 20.8 [15.1 to 26.5]
  At Week 38 | 17.6 [12.7 to 22.6] | 15.7 [11.2 to 20.3] | 14.7 [9.8 to 19.7]
  At Week 42 | 17.2 [12.3 to 22.1] | 18.5 [13.7 to 23.4] | 18.3 [12.9 to 23.7]
  At Week 46 | 15.0 [10.3 to 19.6] | 18.5 [13.7 to 23.4] | 14.7 [9.8 to 19.7]
  At Week 50 | 22.0 [16.6 to 27.4] | 23.0 [17.7 to 28.2] | 18.3 [12.9 to 23.7]
  At Week 54 | 18.1 [13.1 to 23.1] | 14.9 [10.5 to 19.4] | 15.7 [10.7 to 20.8]
  At Week 58 | 18.9 [13.8 to 24.0] | 19.8 [14.8 to 24.7] | 16.2 [11.1 to 21.4]
  At Week 62 | 17.2 [12.3 to 22.1] | 18.5 [13.7 to 23.4] | 13.2 [8.5 to 17.9]

18. Secondary Outcome: Stage 1: Percentage of Participants Who Achieved >=70% American College of Rheumatology (ACR70) Response Using ESR
Description: ACR70-ESR was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 50% improvement from baseline in the tender/painful joint count. ii) A 70% improvement from baseline in the swollen joint count. iii) A 70% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS)(0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3, with lower scores meaning less disability, e) ESR.
Time Frame: At Weeks 2, 6, 14, 18, 22
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
percentage of participants
  At Week 2 | 0.9 [0.0 to 2.1] | 1.1 [0.1 to 2.1]
  At Week 6 | 5.7 [2.7 to 8.7] | 6.1 [3.8 to 8.3]
  At Week 14 | 9.7 [5.8 to 13.5] | 7.4 [5.0 to 9.8]
  At Week 18 | 14.5 [10.0 to 19.1] | 11.0 [8.1 to 13.9]
  At Week 22 | 11.0 [6.9 to 15.1] | 11.2 [8.3 to 14.1]

19. Secondary Outcome: Stage 2 and 3: Percentage of Participants Who Achieved >=70% American College of Rheumatology (ACR70) Response Using ESR
Description: ACR70-ESR was defined as a dichotomous variable, for which a participant was defined as either a responder or a non-responder. Participant was defined as a responder if all of the following criteria are met: i) A 50% improvement from baseline in the tender/painful joint count. ii) A 70% improvement from baseline in the swollen joint count. iii) A 70% improvement from baseline in at least 3 of the following 5 variables: a) Participant global assessment of disease activity (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), b) Physician global assessment of disease activity (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), c) Participant pain assessment (VAS) (0=very good, no symptoms;100=very poor, severe symptoms), d) HAQ-DI, total score ranged from 0-3, with lower scores meaning less disability, e) ESR.
Time Frame: At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 248 | 197
percentage of participants
  At Week 26 | 15.4 [10.7 to 20.1] | 15.3 [10.8 to 19.8] | 12.7 [8.0 to 17.3]
  At Week 30 | 15.4 [10.7 to 20.1] | 14.1 [9.8 to 18.4] | 11.7 [7.2 to 16.2]
  At Week 34 | 16.7 [11.9 to 21.6] | 16.9 [12.3 to 21.6] | 19.3 [13.8 to 24.8]
  At Week 38 | 16.3 [11.5 to 21.1] | 16.1 [11.6 to 20.7] | 14.2 [9.3 to 19.1]
  At Week 42 | 14.5 [10.0 to 19.1] | 17.3 [12.6 to 22.1] | 15.7 [10.7 to 20.8]
  At Week 46 | 15.4 [10.7 to 20.1] | 16.9 [12.3 to 21.6] | 13.2 [8.5 to 17.9]
  At Week 50 | 20.7 [15.4 to 26.0] | 22.6 [17.4 to 27.8] | 15.7 [10.7 to 20.8]
  At Week 54 | 17.2 [12.3 to 22.1] | 13.3 [9.1 to 17.5] | 13.7 [8.9 to 18.5]
  At Week 58 | 17.2 [12.3 to 22.1] | 18.1 [13.3 to 22.9] | 14.7 [9.8 to 19.7]
  At Week 62 | 16.3 [11.5 to 21.1] | 18.1 [13.3 to 22.9] | 15.2 [10.2 to 20.2]

20. Secondary Outcome: Stage 1: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Weeks 2, 6, 14, 18, and 22
Description: The HAQ-DI score was defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled), where lower scores indicated less disability. Negative change from baseline indicates improvement (less disability).
Time Frame: Baseline, Weeks 2, 6, 14, 18, and 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
score on a scale
  Baseline: number analyzed (Participants) | 227 | 443
  Baseline | 1.32 (0.55) | 1.34 (0.58)
  Change at Week 2: number analyzed (Participants) | 222 | 435
  Change at Week 2 | -0.21 (0.42) | -0.28 (0.45)
  Change at Week 6: number analyzed (Participants) | 223 | 438
  Change at Week 6 | -0.33 (0.50) | -0.37 (0.53)
  Change at Week 14: number analyzed (Participants) | 215 | 412
  Change at Week 14 | -0.35 (0.55) | -0.35 (0.54)
  Change at Week 18: number analyzed (Participants) | 213 | 404
  Change at Week 18 | -0.41 (0.53) | -0.43 (0.58)
  Change at Week 22: number analyzed (Participants) | 216 | 399
  Change at Week 22 | -0.35 (0.59) | -0.39 (0.59)

21. Secondary Outcome: Stage 2 and 3: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Description: as for outcome 20
Time Frame: Baseline, Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 249 | 197
score on a scale
  Change at Week 26: number analyzed (Participants) | 212 | 195 | 192
  Change at Week 26 | -0.40 (0.59) | -0.44 (0.63) | -0.40 (0.58)
  Change at Week 30: number analyzed (Participants) | 203 | 187 | 186
  Change at Week 30 | -0.40 (0.57) | -0.46 (0.62) | -0.38 (0.59)
  Change at Week 34: number analyzed (Participants) | 199 | 180 | 182
  Change at Week 34 | -0.47 (0.58) | -0.50 (0.61) | -0.44 (0.58)
  Change at Week 38: number analyzed (Participants) | 188 | 181 | 171
  Change at Week 38 | -0.43 (0.59) | -0.46 (0.61) | -0.41 (0.63)
  Change at Week 42: number analyzed (Participants) | 180 | 179 | 168
  Change at Week 42 | -0.48 (0.56) | -0.52 (0.65) | -0.46 (0.62)
  Change at Week 46: number analyzed (Participants) | 173 | 174 | 163
  Change at Week 46 | -0.48 (0.60) | -0.51 (0.67) | -0.43 (0.60)
  Change at Week 50: number analyzed (Participants) | 174 | 170 | 160
  Change at Week 50 | -0.49 (0.58) | -0.55 (0.64) | -0.47 (0.61)
  Change at Week 54: number analyzed (Participants) | 167 | 163 | 160
  Change at Week 54 | -0.49 (0.58) | -0.49 (0.64) | -0.39 (0.63)
  Change at Week 58: number analyzed (Participants) | 165 | 160 | 152
  Change at Week 58 | -0.49 (0.59) | -0.52 (0.64) | -0.44 (0.60)
  Change at Week 62: number analyzed (Participants) | 162 | 160 | 154
  Change at Week 62 | -0.47 (0.59) | -0.51 (0.64) | -0.42 (0.61)

22. Secondary Outcome: Stage 1: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Scores at Weeks 2, 6, 14, 18, and 22
Description: Disease activity was assessed using RAPID3, based on participant-reported multi-dimensional health assessment questionnaire (MDHAQ). RAPID3 included 3 core data set measures of physical function, pain, and participant global estimate.Physical function=mean of scores from 10 individual questions on activities of daily living (each question scored from '0'=no difficulty to '3'=much difficulty), scores were transformed to give total score=0-10, higher scores=greater difficulty.Pain and global estimate of health measured on Likert scale from '0'=no pain to '10'=pain as bad as it could be. RAPID3 composite score: mean of physical function, pain, and global assessment scores, ranging from 0 to 10, higher values=greater disease activity. Total score range of RAPID3 score was 0=no difficulty; 30=greater difficultly, and disease activity categories were as follows: remission: 0-3, low: >3.1 to 6, moderate: >6.1-12, and high: >12.1. Negative change from baseline indicates less disease activity.
Time Frame: Baseline, Weeks 2, 6, 14, 18, and 22
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
score on a scale
  Baseline: number analyzed (Participants) | 224 | 438
  Baseline | 17.03 (4.76) | 17.37 (4.76)
  Change at Week 2: number analyzed (Participants) | 219 | 432
  Change at Week 2 | -2.99 (4.42) | -3.79 (4.89)
  Change at Week 6: number analyzed (Participants) | 220 | 430
  Change at Week 6 | -4.15 (5.14) | -5.05 (5.62)
  Change at Week 14: number analyzed (Participants) | 213 | 400
  Change at Week 14 | -5.04 (5.80) | -4.91 (6.47)
  Change at Week 18: number analyzed (Participants) | 213 | 402
  Change at Week 18 | -5.99 (5.96) | -5.73 (6.51)
  Change at Week 22: number analyzed (Participants) | 212 | 391
  Change at Week 22 | -4.71 (6.42) | -5.41 (6.54)

23. Secondary Outcome: Stage 2 and 3: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Scores At Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Description: Disease activity was assessed using RAPID3, based on participant-reported multi-dimensional health assessment questionnaire (MDHAQ). RAPID3 included 3 core data set measures of physical function, pain and participant global estimate. Physical function=mean of scores from 10 individual questions on activities of daily living (each question scored from '0'=no difficulty to '3'=much difficulty), scores were transformed to give total score=0-10, higher scores=greater difficulty. Pain and global estimate of health measured on Likert scale from '0'=no pain to '10'=pain as bad as it could be. RAPID3 composite score: mean of physical function, pain, and global assessment scores, ranging from 0 to 10, higher values=greater disease activity. Total score range of RAPID3 score was 0=no difficulty-30=greater difficultly, and disease activity categories were as follows: remission: 0-3, low: >3.1 to 6, moderate: >6.1-12, and high: >12.1. Negative change from baseline indicates less disease activity.
Time Frame: Baseline, Weeks 26, 30, 34, 38, 42, 46, 50, 54, 58, and 62
Population: The FAS population included all participants who received at least 1 dose of study drug and had at least 1 post-baseline RAPID3 efficacy assessment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 249 | 197
score on a scale
  Change at Week 26: number analyzed (Participants) | 209 | 183 | 191
  Change at Week 26 | -5.81 (6.23) | -6.34 (6.55) | -5.64 (6.43)
  Change at Week 30: number analyzed (Participants) | 199 | 181 | 185
  Change at Week 30 | -5.43 (6.38) | -6.41 (6.81) | -5.26 (6.67)
  Change at Week 34: number analyzed (Participants) | 194 | 176 | 179
  Change at Week 34 | -6.24 (6.06) | -7.39 (6.51) | -6.22 (6.75)
  Change at Week 38: number analyzed (Participants) | 183 | 177 | 170
  Change at Week 38 | -5.91 (6.25) | -6.59 (7.14) | -5.86 (6.94)
  Change at Week 42: number analyzed (Participants) | 175 | 173 | 164
  Change at Week 42 | -6.69 (6.10) | -7.40 (6.82) | -6.49 (6.49)
  Change at Week 46: number analyzed (Participants) | 174 | 170 | 162
  Change at Week 46 | -6.34 (6.35) | -7.11 (6.99) | -5.79 (6.53)
  Change at Week 50: number analyzed (Participants) | 167 | 162 | 160
  Change at Week 50 | -6.85 (6.36) | -7.94 (7.22) | -6.48 (6.63)
  Change at Week 54: number analyzed (Participants) | 163 | 160 | 157
  Change at Week 54 | -6.63 (6.33) | -7.11 (7.27) | -5.38 (6.64)
  Change at Week 58: number analyzed (Participants) | 162 | 156 | 152
  Change at Week 58 | -6.84 (6.54) | -7.83 (7.05) | -6.41 (6.25)
  Change at Week 62: number analyzed (Participants) | 204 | 183 | 184
  Change at Week 62 | -5.35 (6.83) | -6.28 (7.46) | -5.74 (6.67)

24. Secondary Outcome: Stage 1: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Total Score at Weeks 14 and 22
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental heallth) with a Subscale Total score for each scaled from 0 (minimum) to 100 (maximum) with a Total Overall score on a 0-800 scale, with higher scores indicating better health. where higher score indicates highest level of functioning. These 8 aspects can also be summarized as Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life). A positive change indicates improvement while a negative change indicates worsening of health status and quality of life. Change from baseline in overall total score for SF-36 was reported in this outcome measure.
Time Frame: Baseline, Weeks 14 and 22
Population: The ITT population included all participants who were randomized. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
score on a scale
  Baseline: number analyzed (Participants) | 223 | 437
  Baseline | 360.46 (116.64) | 358.20 (126.93)
  Change at Week 14: number analyzed (Participants) | 212 | 399
  Change at Week 14 | 79.90 (124.86) | 77.59 (124.72)
  Change at Week 22: number analyzed (Participants) | 211 | 390
  Change at Week 22 | 90.02 (122.36) | 82.94 (129.28)

25. Secondary Outcome: Stage 2 and 3: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Total Score at Weeks 38 and 62
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental heallth) with a Subscale Total score for each scaled from 0 (minimum) to 100 (maximum) with a Total Overall score on a 0-800 scale, with higher scores indicating better health. where higher score indicates highest level of functioning. Total score for each subscale scaled from 0 (minimum) to 100 (maximum), where higher score indicates highest level of functioning. These 8 aspects can also be summarized as PCS with score range 0-100 (higher score-better quality of life) and a MCS with score range 0-100 (higher score-better quality of life). A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline, Weeks 38 and 62
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 249 | 197
score on a scale
  Change at Week 38: number analyzed (Participants) | 182 | 176 | 169
  Change at Week 38 | 95.10 (127.26) | 96.93 (136.80) | 87.61 (129.67)
  Change at Week 62: number analyzed (Participants) | 203 | 213 | 182
  Change at Week 62 | 81.56 (143.91) | 95.24 (148.23) | 87.51 (122.36)

26. Secondary Outcome: Stage 1: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Score for Physical and Mental Components at Weeks 14 and 22
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. A Subscale Total score for each scaled from 0 (minimum) to 100 (maximum). Total score for each subscale scaled from 0 (minimum) to 100 (maximum), where higher score indicates highest level of functioning. These 2 subscale aspects can also be summarized as PCS with score range 0-100 (higher score-better quality of life) and a MCS with score range 0-100 (higher score-better quality of life). A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline, Weeks 14 and 22
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 446
score on a scale
  Baseline (Physical Component): number analyzed (Participants) | 223 | 437
  Baseline (Physical Component) | 30.22 (7.72) | 30.53 (7.24)
  Change at Week 14 (Physical Component): number analyzed (Participants) | 212 | 399
  Change at Week 14 (Physical Component) | 5.42 (7.86) | 5.64 (8.82)
  Change at Week 22 (Physical Component): number analyzed (Participants) | 211 | 390
  Change at Week 22 (Physical Component) | 5.61 (8.36) | 6.03 (8.79)
  Baseline (Mental Component): number analyzed (Participants) | 223 | 437
  Baseline (Mental Component) | 43.59 (11.57) | 43.02 (12.45)
  Change at Week 14 (Mental Component): number analyzed (Participants) | 212 | 399
  Change at Week 14 (Mental Component) | 3.05 (10.36) | 2.56 (10.38)
  Change at Week 22 (Mental Component): number analyzed (Participants) | 211 | 390
  Change at Week 22 (Mental Component) | 4.05 (9.48) | 2.71 (10.83)

27. Secondary Outcome: Stage 2 and 3: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Score for Physical and Mental Components at Weeks 38 and 62
Description: as for outcome 26
Time Frame: Baseline, Weeks 38 and 62
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 249 | 197
score on a scale
  Change at Week 38 (Physical Component): number analyzed (Participants) | 182 | 176 | 169
  Change at Week 38 (Physical Component) | 6.94 (8.37) | 6.86 (9.31) | 6.22 (9.62)
  Change at Week 62 (Physical Component): number analyzed (Participants) | 203 | 213 | 182
  Change at Week 62 (Physical Component) | 6.14 (8.79) | 6.23 (9.78) | 6.11 (8.60)
  Change at Week 38 (Mental Component): number analyzed (Participants) | 182 | 176 | 169
  Change at Week 38 (Mental Component) | 3.09 (10.55) | 3.38 (11.32) | 3.10 (10.58)
  Change at Week 62 (Mental Component): number analyzed (Participants) | 203 | 213 | 182
  Change at Week 62 (Mental Component) | 2.45 (10.92) | 3.93 (11.59) | 3.16 (10.29)

28. Secondary Outcome: Stage 2 and 3: Minimum Observed Serum Concentration (Cmin) of NI-071 and Remicade US
Description: Drug concentrations in blood were evaluated from week 46 to week 54 after the initial administration date.
  Blood sampling was performed before administration of week 46, at the end of the infusion, and at 4 hours, 24 hours, 7 days (week 47), 14 days (week 48), 28 days (week 50), and 56 days (before administration of week 54). Cmin was define as the lowest drug concentration among all blood sampling points for an individual patient.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 159 | 155 | 146
ng/mL | 839.1 (1322.2) | 754.1 (1380.0) | 762.6 (1207.2)

29. Secondary Outcome: Stage 2 and 3: Time to Reach the Maximum Serum Concentration (Tmax) of NI-071 and Remicade US
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 159 | 155 | 146
hours | 52.37 (243.64) | 41.57 (217.28) | 32.98 (191.02)

30. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical condition that occurs in participants while participating in a clinical study and does not necessarily have a causal relationship with the use of the study treatment. A TEAE was defined as an adverse event with a start date on or after the first dose of Investigational product (IP), or a start date before the date of the first dose of IP but increased in severity on or after the date of the first dose of IP. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Number of participants with TEAEs and Serious TEAEs were reported.
Time Frame: Baseline up to Week 62
Population: The safety population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Stages 1, 2 and 3: NI-071 Group: Participants received IV infusion of NI-071 at a dose of 3 milligrams/kilograms (mg/kg) at Weeks 0, 2, 6, 14 during stage 1 and at Weeks 22, 30, 38, 46, and 54 during stage 2. Participants were followed up to Week 62 (Stage 3).
- Stage 2 and Stage 3: Remicade US to Remicade-US Group: Participants who received Remicade US during stage 1 and were re-randomized during stage 2 to continue Remicade-US dose 3 mg/kg from Week 22 through Week 54 with every 8 weeks dosing intervals. Participants were followed up to Week 62 (Stage 3).
- Stage 2 and Stage 3: Remicade US to Switch Group: Participants who received Remicade US during stage 1 and were re-randomized during stage 2 received IV infusion of NI-071 at Week 22 followed by Remicade-US at Week 30, followed by NI-071 at Weeks 38, 46, and 54. Participants were followed up to week 62 (Stage 3).
Arm/Group | Stages 1, 2 and 3: NI-071 Group | Stage 1: Remicade-US Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 451 | 254 | 197
Participants
  Participants with TEAEs | 157 | 330 | 181 | 149
  Participants with Serious TEAEs | 19 | 41 | 28 | 13

31. Secondary Outcome: Number of Participants With TEAEs of Special Interest
Description: A TEAE was defined as an adverse event with a start date on or after the first dose of IP or a start date before the date of the first dose of IP but increased in severity on or after the date of the first dose of IP.
Time Frame: Baseline up to Week 62
Population: The safety population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1, Stage 2, and Stage 3: NI-071 Group: Participants received IV infusion of NI-071 at a dose of 3 mg/kg at Weeks 0, 2, 6, 14 during stage 1 and at Weeks 22, 30, 38, 46, and 54 during stage 2. Participants were followed up to Week 62 (Stage 3).
Arm/Group | Stage 1, Stage 2, and Stage 3: NI-071 Group | Stage 1: Remicade-US Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 451 | 254 | 197
Participants | 33 | 68 | 43 | 25

32. Secondary Outcome: Stage 1: Number of Participants With Positive Serum Anti-drug Antibodies (ADA)
Description: Number of Participants With Positive Serum ADA are reported.
Time Frame: Baseline, Weeks 2, 6, 14, and 22
Population: The safety population included participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specific time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 451
Participants
  Baseline: number analyzed (Participants) | 222 | 447
  Baseline | 2 | 15
  At Week 2: number analyzed (Participants) | 226 | 439
  At Week 2 | 18 | 44
  At Week 6: number analyzed (Participants) | 223 | 437
  At Week 6 | 59 | 143
  At Week 14: number analyzed (Participants) | 215 | 412
  At Week 14 | 150 | 303
  At Week 22: number analyzed (Participants) | 213 | 396
  At Week 22 | 187 | 337

33. Secondary Outcome: Stage 2 and 3: Number of Participants With Positive Serum Anti-drug Antibodies (ADA)
Description: Number of Participants With Positive Serum Anti-drug Antibodies (ADA) are reported.
Time Frame: At Weeks 30, 38, 46, 54, and 62
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 254 | 197
Participants
  At Week 30: number analyzed (Participants) | 201 | 185 | 185
  At Week 30 | 185 | 166 | 164
  At Week 38: number analyzed (Participants) | 183 | 181 | 169
  At Week 38 | 167 | 162 | 146
  At Week 46: number analyzed (Participants) | 173 | 172 | 161
  At Week 46 | 153 | 150 | 141
  At Week 54: number analyzed (Participants) | 162 | 163 | 158
  At Week 54 | 147 | 145 | 141
  At Week 62: number analyzed (Participants) | 208 | 217 | 184
  At Week 62 | 187 | 191 | 165

34. Secondary Outcome: Stage 1: Number of Participants With Positive Serum Neutralizing Antibodies
Description: Number of Participants with Positive Serum neutralizing Antibodies were reported.
Time Frame: Baseline, Weeks 2, 6, 14, and 22
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: NI-071 Group | Stage 1: Remicade-US Group
Number analyzed (Participants) | 227 | 451
Participants
  Baseline: number analyzed (Participants) | 2 | 15
  Baseline | 1 | 7
  At Week 2: number analyzed (Participants) | 18 | 44
  At Week 2 | 1 | 10
  At Week 6: number analyzed (Participants) | 59 | 153
  At Week 6 | 11 | 34
  At Week 14: number analyzed (Participants) | 150 | 303
  At Week 14 | 53 | 122
  At Week 22: number analyzed (Participants) | 187 | 337
  At Week 22 | 80 | 143

35. Secondary Outcome: Stage 2 and 3: Number of Participants With Positive Serum Neutralizing Antibodies
Description: Number of Participants with Positive Serum neutralizing Antibodies were reported.
Time Frame: At Weeks 30, 38, 46, 54, and 62
Population: The safety population included participants who received at least 1 dose of study drug. Here, "Number Analyzed" signifies those participants who were evaluable at specific time point. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 and Stage 3: NI-071 Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
Number analyzed (Participants) | 227 | 254 | 197
Participants
  At Week 30: number analyzed (Participants) | 185 | 166 | 164
  At Week 30 | 92 | 90 | 78
  At Week 38: number analyzed (Participants) | 167 | 162 | 146
  At Week 38 | 94 | 96 | 69
  At Week 46: number analyzed (Participants) | 153 | 150 | 141
  At Week 46 | 78 | 87 | 75
  At Week 54: number analyzed (Participants) | 147 | 145 | 141
  At Week 54 | 77 | 87 | 75
  At Week 62: number analyzed (Participants) | 187 | 191 | 165
  At Week 62 | 114 | 124 | 97

ADVERSE EVENTS:
Time Frame: Baseline up to Week 62
Description: The safety population included participants who received at least 1 dose of study drug at Baseline. The analyses were calculated by the number of All-Cause Mortality/safety population, the number of SAE's/safety population and the number of oher AE's/safety population. The patient number of safety population is the number of patients evaluated at baseline, which is different from the number of patients who started to Stage 2 or 3.
Groups:
- Stage 1, 2 and 3: NI-071 Group: Participants received IV infusion of NI-071 at a dose of 3 mg/kg at Weeks 0, 2, 6, 14 during stage 1 and at Weeks 22, 30, 38, 46, and 54 during stage 2. Participants were followed up to Week 62 (Stage 3).
Arm/Group | Stage 1, 2 and 3: NI-071 Group | Stage 1: Remicade-US Group | Stage 2 and Stage 3: Remicade US to Remicade-US Group | Stage 2 and Stage 3: Remicade US to Switch Group
All-Cause Mortality (participants affected / at risk) | 1/227 | 1/451 | 0/254 | 0/197
Serious Adverse Events (participants affected / at risk) | 19/227 | 41/451 | 28/254 | 13/197
Other Adverse Events (participants affected / at risk) | 96/227 | 174/451 | 80/254 | 94/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1, 2 and 3: NI-071 Group (N=227) | Stage 1: Remicade-US Group (N=451) | Stage 2 and Stage 3: Remicade US to Remicade-US Group (N=254) | Stage 2 and Stage 3: Remicade US to Switch Group (N=197)
Abdominal abscess (Infections and infestations) | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 2 | 1 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 1
Squamous cell carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 3 | 3 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Autoimmune encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Hysterectomy (Surgical and medical procedures) | 0 | 1 | 0 | 1
Medical device removal (Surgical and medical procedures) | 0 | 1 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1, 2 and 3: NI-071 Group (N=227) | Stage 1: Remicade-US Group (N=451) | Stage 2 and Stage 3: Remicade US to Remicade-US Group (N=254) | Stage 2 and Stage 3: Remicade US to Switch Group (N=197)
Bronchitis (Infections and infestations) | 13 | 16 | 10 | 6
Nasopharyngitis (Infections and infestations) | 28 | 43 | 22 | 21
Upper Respiratory Tract Infection (Infections and infestations) | 24 | 41 | 21 | 20
Headache (Nervous system disorders) | 16 | 21 | 8 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 16 | 6 | 10
Alanine Aminotransferase Increased (Investigations) | 8 | 21 | 8 | 13
Aspartate Aminotransferase Increased (Investigations) | 4 | 16 | 5 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT02990806/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT02990806/SAP_001.pdf